CLINICAL TRIAL: NCT02632526
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD5718 After Single and Multiple Ascending Dose Administration to Healthy Male Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD5718 After Single and Multiple Ascending Dose Administration to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D7550C00001
Record Dates: First submitted 2015-12-07; First posted 2015-12-16 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Healthy Male Subjects; Cardiovascular Disease
Keywords: AZD5718 oral suspension crystalline; AZD5718 oral suspension amorphous; Single ascending dose/multiple ascending dose (SAD/MAD); Placebo-controlled; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (17):
- AZD5718 amorphous form, treatment 1 (Part A) (Experimental): Starting dose 25 mg/day, single ascending dose
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 2 (Part A) (Experimental): Single dose of AZD5718 amorphous suspension
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 3 (Part A) (Experimental): Single dose of AZD5718 amorphous suspension
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 4 (Part A) (Experimental): Single dose of AZD5718 amorphous suspension
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 5 (Part A) (Experimental): Single dose of AZD5718 amorphous suspension
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 6 (Part A) (Experimental): Single dose of AZD5718 amorphous suspension
  Interventions: Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718, crystalline form, treatment 7 (Part A) (Experimental): Crystalline suspension (Part A), dosage lower than highest dose used with amorphous suspension, single ascending dose
  Interventions: Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 crystalline form, treatment 8 (Part A) (Experimental): Crystalline suspension (Part A), dosage lower than highest dose used with amorphous suspension, single ascending dose
  Interventions: Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous form, treatment 1 (Part B) (Experimental): Once or twice daily from Days 2 to 9 and single doses on Days 1 and 10, dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)
- AZD5718 amorphous form, treatment 2 (Part B) (Experimental): Once or twice daily from Days 2 to 9 and single doses on Days 1 and 10, dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)
- AZD5718 amorphous form, treatment 3 (Part B) (Experimental): Once or twice daily from Days 2 to 9 and single doses on Days 1 and 10, dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)
- AZD5718 amorphous form, treatment 4 (Part B) (Experimental): Once or twice daily from Days 2 to 9 and single doses on Days 1 and 10, dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)
- AZD5718 amorphous/crystalline form, repeat 1 (Part A) (Experimental): Single dose of AZD5718 amorphous form (Part A) Crystalline form (Part A), dosage lower than highest dose used with amorphous form, single ascending dose
  Interventions: Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A); Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous/crystalline form, repeat 2 (Part A) (Experimental): Single dose of AZD5718 amorphous form (Part A) Crystalline form (Part A), dosage lower than highest dose used with amorphous form, single ascending dose
  Interventions: Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A); Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A); Drug: AZD5718 placebo oral suspension
- AZD5718 amorphous/crystalline, repeat 3 (Part A) (Experimental): Single dose of AZD5718 amorphous form (Part A) Crystalline form (Part A), dosage lower than highest dose used with amorphous form, single ascending dose
  Interventions: Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A); Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A)
- AZD5718 amorphous form, repeat 1 (Part B) (Experimental): Twice daily dosing (Day 1 - 9) and once daily dosing (Day 10), dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)
- AZD5718 amorphous form, repeat 2 (Part B) (Experimental): Twice daily dosing (Day 1 - 9) and once daily dosing (Day 10), dosage TBD (Part A)
  Interventions: Drug: AZD5718 placebo oral suspension; Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B)

INTERVENTIONS:
Drug: AZD5718 oral suspension crystalline form (1 to 100 mg/mL) (Part A) — Oral suspension single dose
  Arms: AZD5718 amorphous/crystalline form, repeat 1 (Part A); AZD5718 amorphous/crystalline form, repeat 2 (Part A); AZD5718 amorphous/crystalline, repeat 3 (Part A); AZD5718 crystalline form, treatment 8 (Part A); AZD5718, crystalline form, treatment 7 (Part A)
Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part A) — Single and multiple doses
  Arms: AZD5718 amorphous form, treatment 1 (Part A); AZD5718 amorphous form, treatment 2 (Part A); AZD5718 amorphous form, treatment 3 (Part A); AZD5718 amorphous form, treatment 4 (Part A); AZD5718 amorphous form, treatment 5 (Part A); AZD5718 amorphous form, treatment 6 (Part A); AZD5718 amorphous/crystalline form, repeat 1 (Part A); AZD5718 amorphous/crystalline form, repeat 2 (Part A); AZD5718 amorphous/crystalline, repeat 3 (Part A)
Drug: AZD5718 placebo oral suspension — Single and multiple doses
  Arms: AZD5718 amorphous form, repeat 1 (Part B); AZD5718 amorphous form, repeat 2 (Part B); AZD5718 amorphous form, treatment 1 (Part A); AZD5718 amorphous form, treatment 1 (Part B); AZD5718 amorphous form, treatment 2 (Part A); AZD5718 amorphous form, treatment 2 (Part B); AZD5718 amorphous form, treatment 3 (Part A); AZD5718 amorphous form, treatment 3 (Part B); AZD5718 amorphous form, treatment 4 (Part A); AZD5718 amorphous form, treatment 4 (Part B); AZD5718 amorphous form, treatment 5 (Part A); AZD5718 amorphous form, treatment 6 (Part A); AZD5718 amorphous/crystalline form, repeat 1 (Part A); AZD5718 amorphous/crystalline form, repeat 2 (Part A); AZD5718 crystalline form, treatment 8 (Part A); AZD5718, crystalline form, treatment 7 (Part A)
Drug: AZD5718 oral suspension amorphous (1 to 100 mg/mL) (Part B) — Single and multiple doses
  Arms: AZD5718 amorphous form, repeat 1 (Part B); AZD5718 amorphous form, repeat 2 (Part B); AZD5718 amorphous form, treatment 1 (Part B); AZD5718 amorphous form, treatment 2 (Part B); AZD5718 amorphous form, treatment 3 (Part B); AZD5718 amorphous form, treatment 4 (Part B)

SUMMARY:
This is a phase I, randomised, single-blind, placebo-controlled, first-in-human (FIH) single and multiple ascending dose study consisting of two parts (Part A [SAD] and Part B [MAD]) to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD5718 in healthy male subjects

DETAILED DESCRIPTION:
This is a phase I, randomised, single-blind, placebo-controlled, first-in-human (FIH) single and multiple ascending dose study consisting of two parts (Part A [SAD] and Part B [MAD]) to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD5718 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male subjects aged 18 - 50 years, inclusive, with suitable veins for cannulation or repeated venepuncture
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive
4. Provision of signed, written and dated informed consent for optional genetic research

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of investigational medicinal product (IMP)
4. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results at screening and check-in, as judged by the investigator, including:

   * Alanine aminotransferase (ALT) > upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) > ULN;
   * Bilirubin (total) > ULN; and
   * Gamma glutamyl transpeptidase (GGT) > ULN
5. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV)
6. Suspicion or known Gilbert's syndrome
7. Abnormal vital signs, after 10 minutes supine rest, at screening and check-in, defined as any of the following:

   * Systolic blood pressure(BP) (SBP) < 90mmHg or ≥ 140 mmHg;
   * Diastolic BP (DBP) < 50mmHg or ≥ 90 mmHg; and
   * Pulse < 45 or > 85 beats per minute (bpm)
8. Any clinically significant abnormalities (at screening and check-in) in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy
9. Prolonged QTcF (QT interval corrected for heart rate using Fridericia's formula) > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome, at screening and check-in
10. PR(PQ) interval (ECG interval measured from the onset of the P wave to the onset of the QRS complex) shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation), at screening and check-in
11. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation, at screening and check-in
12. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation, at screening and check-in
13. Known or suspected history of drug abuse, as judged by the investigator
14. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening
15. Any history of alcohol abuse or excessive intake of alcohol, as judged by the investigator
16. Positive screen for drugs of abuse, alcohol or cotinine (nicotine) at screening or admission to the unit
17. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718
18. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator
19. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP
20. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the administration of IMP or longer if the medication has a long half-life
21. Plasma donation within 1 month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening
22. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of IMP in this study. The period of exclusion is 3 months after the final dose from a previous study
23. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
24. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives
25. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements
26. Subjects who are vegans or have medical dietary restrictions
27. Subjects who cannot communicate reliably with the investigator

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
28. Previous bone marrow transplant
29. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, FFPM, Principal Investigator — Parexel
Locations (1):
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted on 96 healthy male participants at a single center: PAREXEL Early Phase Clinical Unit - London. This study consisted of 2 parts: Part A - single ascending dose (SAD) and Part B - multiple ascending dose (MAD).
Pre-assignment Details: Screening period was from Day -28 and Day -1. Participants signed informed consent form; demographic data, medical history and concomitant medication details were collected; weight, height and body mass index were measured; inclusion/exclusion criteria were checked, serology and screening of urinary drugs of abuse, alcohol and cotinine were done
Groups:
- Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 in amorphous state at dose levels 25 mg, 50 mg, 100 mg, 300 mg, 600 mg & 1200mg with 6 participants in each dose level
- Part A (Crystalline Suspension): Participants received single dose of oral suspension of AZD5718 in crystalline state at dose levels 100 mg & 300 mg with 6 participants in each dose level
- Part B (Amorphous Suspension): Participants received multiple daily doses of oral suspension of AZD5718 in amorphous state at dose levels 60 mg, 180 mg, 360 mg & 600 mg with 6 participants in each dose level
- Placebo - Part A (Amorphous Suspension): 2 participants per dose level received single dose of placebo in Part A (Amorphous suspension)
- Placebo - Part A (Crystalline Suspension): 2 participants per dose level received single dose of placebo in Part A (Crystalline suspension)
- Placebo - Part B (Amorphous Suspension): 2 participants per dose level received single dose of placebo in Part B (Amorphous suspension)
Period: Overall Study
Arm/Group | Part A (Amorphous Suspension) | Part A (Crystalline Suspension) | Part B (Amorphous Suspension) | Placebo - Part A (Amorphous Suspension) | Placebo - Part A (Crystalline Suspension) | Placebo - Part B (Amorphous Suspension)
Started | 36 | 12 | 24 | 12 | 4 | 8
Completed | 36 | 12 | 24 | 12 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Amorphous Suspension) | Part A (Crystalline Suspension) | Part B (Amorphous Suspension) | Placebo - Part A (Amorphous Suspension) | Placebo - Part A (Crystalline Suspension) | Placebo - Part B (Amorphous Suspension) | Total
Number analyzed (Participants) | 36 | 12 | 24 | 12 | 4 | 8 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The number analyzed in row differs from overall since the data for Part A (Amorphous Suspension), Part A (Crystalline Suspension), Part B (Amorphous Suspension), Placebo - Part A (Amorphous Suspension), Placebo - Part A (Crystalline Suspension), Placebo - Part B (Amorphous Suspension) are presented in different rows.
  Years
    Part A (Amorphous Suspension): number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0 | 36
    Part A (Amorphous Suspension) | 34.3 (8.85) |  |  |  |  |  | 34.3 (8.85)
    Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 12
    Part A (Crystalline Suspension) |  | 33.2 (11.64) |  |  |  |  | 33.2 (11.64)
    Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 24 | 0 | 0 | 0 | 24
    Part B (Amorphous Suspension) |  |  | 35.5 (7.32) |  |  |  | 35.5 (7.32)
    Placebo - Part A (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 12
    Placebo - Part A (Amorphous Suspension) |  |  |  | 34.9 (10.23) |  |  | 34.9 (10.23)
    Placebo - Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Placebo - Part A (Crystalline Suspension) |  |  |  |  | 33.3 (5.62) |  | 33.3 (5.62)
    Placebo - Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Placebo - Part B (Amorphous Suspension) |  |  |  |  |  | 38.3 (5.31) | 38.3 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 36 | 12 | 24 | 12 | 4 | 8 | 96
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 24 | 9 | 20 | 9 | 2 | 5 | 69
  Black or African American | 7 | 1 | 1 | 2 | 1 | 0 | 12
  Asian | 4 | 1 | 3 | 1 | 0 | 2 | 11
  Other: Mixed: Black And White | 1 | 1 | 0 | 0 | 1 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 35 | 11 | 23 | 12 | 3 | 7 | 91
Height [Mean (Standard Deviation); unit: Centimeter] — Population: The number analyzed in row differs from overall since the data for Part A (Amorphous Suspension), Part A (Crystalline Suspension), Part B (Amorphous Suspension), Placebo - Part A (Amorphous Suspension), Placebo - Part A (Crystalline Suspension), Placebo - Part B (Amorphous Suspension) are presented in different rows.
  Centimeter
    Part A (Amorphous Suspension): number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0 | 36
    Part A (Amorphous Suspension) | 179.0 (6.32) |  |  |  |  |  | 179.0 (6.32)
    Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 12
    Part A (Crystalline Suspension) |  | 180.9 (6.95) |  |  |  |  | 180.9 (6.95)
    Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 24 | 0 | 0 | 0 | 24
    Part B (Amorphous Suspension) |  |  | 178.0 (7.07) |  |  |  | 178.0 (7.07)
    Placebo - Part A (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 12
    Placebo - Part A (Amorphous Suspension) |  |  |  | 176.3 (5.33) |  |  | 176.3 (5.33)
    Placebo - Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Placebo - Part A (Crystalline Suspension) |  |  |  |  | 174.3 (3.30) |  | 174.3 (3.30)
    Placebo - Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Placebo - Part B (Amorphous Suspension) |  |  |  |  |  | 175.5 (7.37) | 175.5 (7.37)
Weight [Mean (Standard Deviation); unit: Kilogram] — Population: The number analyzed in row differs from overall since the data for Part A (Amorphous Suspension), Part A (Crystalline Suspension), Part B (Amorphous Suspension), Placebo - Part A (Amorphous Suspension), Placebo - Part A (Crystalline Suspension), Placebo - Part B (Amorphous Suspension) are presented in different rows.
  Kilogram
    Part A (Amorphous Suspension): number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0 | 36
    Part A (Amorphous Suspension) | 79.24 (10.982) |  |  |  |  |  | 79.24 (10.982)
    Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 12
    Part A (Crystalline Suspension) |  | 74.89 (5.450) |  |  |  |  | 74.89 (5.450)
    Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 24 | 0 | 0 | 0 | 24
    Part B (Amorphous Suspension) |  |  | 77.95 (10.369) |  |  |  | 77.95 (10.369)
    Placebo - Part A (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 12
    Placebo - Part A (Amorphous Suspension) |  |  |  | 76.70 (9.547) |  |  | 76.70 (9.547)
    Placebo - Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Placebo - Part A (Crystalline Suspension) |  |  |  |  | 80.50 (2.647) |  | 80.50 (2.647)
    Placebo - Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Placebo - Part B (Amorphous Suspension) |  |  |  |  |  | 74.34 (5.532) | 74.34 (5.532)
Body mass index (BMI) [Mean (Standard Deviation); unit: Kilogram/square meter] — Population: The number analyzed in row differs from overall since the data for Part A (Amorphous Suspension), Part A (Crystalline Suspension), Part B (Amorphous Suspension), Placebo - Part A (Amorphous Suspension), Placebo - Part A (Crystalline Suspension), Placebo - Part B (Amorphous Suspension) are presented in different rows.
  Kilogram/square meter
    Part A (Amorphous Suspension): number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0 | 36
    Part A (Amorphous Suspension) | 24.71 (3.014) |  |  |  |  |  | 24.71 (3.014)
    Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 12
    Part A (Crystalline Suspension) |  | 22.94 (2.265) |  |  |  |  | 22.94 (2.265)
    Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 24 | 0 | 0 | 0 | 24
    Part B (Amorphous Suspension) |  |  | 24.56 (2.456) |  |  |  | 24.56 (2.456)
    Placebo - Part A (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 12
    Placebo - Part A (Amorphous Suspension) |  |  |  | 24.68 (2.764) |  |  | 24.68 (2.764)
    Placebo - Part A (Crystalline Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Placebo - Part A (Crystalline Suspension) |  |  |  |  | 26.55 (1.634) |  | 26.55 (1.634)
    Placebo - Part B (Amorphous Suspension): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Placebo - Part B (Amorphous Suspension) |  |  |  |  |  | 24.14 (1.133) | 24.14 (1.133)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD5718 by Assessment of the Number of Participants With Adverse Events Following Oral Administration of SAD (Part A) and MAD (Part B).
Description: To assess the safety and tolerability of AZD5718 following oral administration of SAD (Part A) and MAD (Part B).
Time Frame: From screening to last followup visit (7-10 days after last dose), up to 6 weeks (Part A) and up to 8 weeks (Part B)
Population: All randomized subjects who received at least 1 dose of IMP and for whom any safety post-dose data were available were included in the safety analysis for the study.
Measure: Number; unit: Participants
Arm/Group | Part A (Amorphous Suspension) | Part A (Crystalline Suspension) | Part B (Amorphous Suspension) | Placebo - Part A (Amorphous Suspension) | Placebo - Part A (Crystalline Suspension) | Placebo - Part B (Amorphous Suspension)
Number analyzed (Participants) | 36 | 12 | 24 | 12 | 4 | 8
Participants
  Any AE | 15 | 2 | 10 | 1 | 1 | 4
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IMP | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Area Under the Plasma Concentration-curve From Time Zero Extrapolated to Infinity (AUC) for Part A - Amorphous and Crystalline Suspension
Description: To assess area under the concentration-time curve from time zero extrapolated to infinity and was estimated by AUC(0-last) + Clast/λz (Clast - the last observed quantifiable concentration) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: At post-dose (Days 1 to 3); 0.5, 1, 2, 3, 4, 6, 8, 24, 36 and 48 hours post-dose and folow up (Day 4 - 72 hours post-dose) (Part A only)
Population: All subjects in the safety analysis set for whom at least one dose of AZD5718 and who had evaluable PK data, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Groups:
- 25 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 25 mg in amorphous state
- 50 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 50 mg in amorphous state
- 100 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 100 mg in amorphous state
- 300 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 300 mg in amorphous state
- 600 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 600 mg in amorphous state
- 1200 mg - Part A (Amorphous Suspension): Participants received single dose of oral suspension of AZD5718 1200 mg in amorphous state
- 100 mg - Part A (Crystalline Suspension): Participants received single dose of oral suspension of AZD5718 100 mg in crystalline state
- 300 mg - Part A (Crystalline Suspension): Participants received single dose of oral suspension of AZD5718 300 mg in crystalline state.
  Presented only based on 5 subjects data.
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*nmol/L | 376.3 (38.09) | 727.0 (15.39) | 1441 (45.26) | 8462 (20.05) | 18810 (42.09) | 35840 (33.71) | 706.7 (24.24) | 1006 (43.72)
Statistical Analysis 1: Comparison: 25 mg - Part A (Amorphous Suspension) vs 50 mg - Part A (Amorphous Suspension) vs 100 mg - Part A (Amorphous Suspension) vs 300 mg - Part A (Amorphous Suspension) vs 600 mg - Part A (Amorphous Suspension) vs 1200 mg - Part A (Amorphous Suspension); Test type: Superiority or Other; Slope = 1.24, 90% CI 2-sided [1.17 to 1.31], Standard Error of Mean 0.0433
Statistical Analysis 2: Comparison: 100 mg - Part A (Crystalline Suspension) vs 300 mg - Part A (Crystalline Suspension); Test type: Superiority or Other; Slope = 0.322, 90% CI 2-sided [-0.0124 to 0.656], Standard Error of Mean 0.182

3. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC) for Part B - Amorphous Suspension
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of the area under plasma concentration-time curve from time zero extrapolated to infinity (AUC) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1 of Part B
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Groups:
- 60 mg - Part B (Amorphous Suspension): Participants received multiple doses of oral suspension of AZD5718 60 mg in amorphous state in 6 cohorts
- 180 mg - Part B (Amorphous Suspension): Participants received multiple doses of oral suspension of AZD5718 180 mg in amorphous state in 6 cohorts
- 360 mg - Part B (Amorphous Suspension): Participants received multiple doses of oral suspension of AZD5718 360 mg in amorphous state in 6 cohorts
- 600 mg - Part B (Amorphous Suspension): Participants received multiple doses of oral suspension of AZD5718 600 mg in amorphous state in 6 cohorts
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*nmol/L | 1087 (24.01) | 3834 (40.94) | 10720 (28.80) | 17010 (47.74)
Statistical Analysis 1: Comparison: 60 mg - Part B (Amorphous Suspension) vs 180 mg - Part B (Amorphous Suspension) vs 360 mg - Part B (Amorphous Suspension) vs 600 mg - Part B (Amorphous Suspension); Day 1; Test type: Superiority or Other; Slope = 1.22, 90% CI 2-sided [1.08 to 1.36], Standard Error of Mean 0.0813

4. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Area Under the Plasma Concentration-curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-last)) for Part A - Amorphous and Crystalline Suspension
Description: To assess area under the area under the plasma concentration-curve from time zero to the time of last quantifiable concentration (AUC(0-last)) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*nmol/L | 264.5 (87.15) | 701.5 (15.83) | 1408 (47.23) | 8395 (20.61) | 18740 (42.13) | 35760 (33.81) | 642.9 (21.55) | 933.2 (41.61)

5. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Area Under the Plasma Concentration-curve Over the Dosing Interval (AUC(0-τ)) for Part B - Amorphous Suspension
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of the area under the plasma concentration-curve over the dosing interval (AUC(0-τ)) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1, Day 9 and Day 10 of Part B
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*nmol/L
  Day 1 | 1018 (22.40) | 3732 (41.19) | 10350 (28.84) | 16290 (48.56)
  Day 9 | 1441 (24.92) | 3312 (33.26) | 13790 (20.56) | 24890 (44.20)
  Day 10 | 1386 (27.40) | 5128 (46.90) | 12760 (31.00) | 23170 (47.49)
Statistical Analysis 1: Comparison: 60 mg - Part B (Amorphous Suspension) vs 180 mg - Part B (Amorphous Suspension) vs 360 mg - Part B (Amorphous Suspension) vs 600 mg - Part B (Amorphous Suspension); Day 10; Test type: Superiority or Other; Slope = 1.23, 90% CI 2-sided [1.08 to 1.38], Standard Error of Mean 0.0851

6. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Observed Maximum Plasma Concentration (Cmax) for Part A - Amorphous and Crystalline Suspension
Description: To assess observed maximum plasma concentration (Cmax) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L | 27.14 (75.96) | 81.62 (36.39) | 170.3 (54.86) | 2358 (32.89) | 5052 (45.82) | 6875 (34.94) | 54.62 (28.35) | 80.24 (39.73)
Statistical Analysis 1: Comparison: 25 mg - Part A (Amorphous Suspension) vs 100 mg - Part A (Amorphous Suspension) vs 300 mg - Part A (Amorphous Suspension) vs 600 mg - Part A (Amorphous Suspension) vs 1200 mg - Part A (Amorphous Suspension); Test type: Superiority or Other; Slope = 1.55, 90% CI 2-sided [1.43 to 1.66], Standard Error of Mean 0.0692
Statistical Analysis 2: Comparison: 100 mg - Part A (Crystalline Suspension) vs 300 mg - Part A (Crystalline Suspension); Test type: Superiority or Other; Slope = 0.350, 90% CI 2-sided [0.0315 to 0.669], Standard Error of Mean 0.176

7. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Observed Maximum Plasma Concentration (Cmax) for Part B - Amorphous Suspension
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of the observed maximum plasma concentration (Cmax) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1, Day 9 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
nmol/L
  Day 1 | 167.3 (19.81) | 846.9 (48.00) | 2561 (31.72) | 4933 (47.63)
  Day 9 | 225.4 (31.70) | 349.8 (34.99) | 3372 (22.69) | 5297 (43.52)
  Day 10 | 219.8 (31.93) | 1243 (55.23) | 3209 (40.01) | 5693 (59.95)
Statistical Analysis 1: Comparison: 60 mg - Part B (Amorphous Suspension) vs 180 mg - Part B (Amorphous Suspension) vs 360 mg - Part B (Amorphous Suspension) vs 600 mg - Part B (Amorphous Suspension); For Day 1; Test type: Superiority or Other; Slope = 1.48, 90% CI 2-sided [1.34 to 1.63], Standard Error of Mean 0.0839
Statistical Analysis 2: Comparison: 60 mg - Part B (Amorphous Suspension) vs 180 mg - Part B (Amorphous Suspension) vs 360 mg - Part B (Amorphous Suspension) vs 600 mg - Part B (Amorphous Suspension); Day 10; Test type: Superiority or Other; Slope = 1.43, 90% CI 2-sided [1.25 to 1.60], Standard Error of Mean 0.104

8. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Time to Reach the Observed Maximum Plasma Concentration (Tmax) for Part A - Amorphous and Crystalline Suspension
Description: To assess the time to reach the observed maximum plasma concentration (tmax) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 2.99 (75.96) [1.00 to 5.98] | 1.02 (36.39) [1.00 to 2.98] | 1.00 (54.86) [0.50 to 3.03] | 1.00 (32.89) [0.52 to 1.00] | 1.00 (45.82) [0.98 to 2.00] | 1.51 (34.94) [1.00 to 2.00] | 3.00 (28.35) [1.00 to 4.00] | 1.98 (39.73) [1.00 to 5.98]

9. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Time to Reach the Observed Maximum Plasma Concentration (Tmax) for Part B - Amorphous Suspension
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of the time to reach the observed maximum plasma concentration (tmax) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1, Day 9 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours
  Day 1 | 0.76 [0.50 to 2.00] | 1.00 [1.00 to 1.00] | 1.01 [1.00 to 2.00] | 1.00 [0.98 to 1.00]
  Day 9 | 1.00 [0.50 to 3.00] | 3.51 [2.00 to 6.02] | 0.99 [0.50 to 1.00] | 2.00 [1.00 to 2.00]
  Day 10 | 0.50 [0.50 to 1.02] | 1.00 [0.98 to 1.02] | 1.00 [1.00 to 1.00] | 1.49 [1.00 to 3.00]

10. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Half-life Associated With Terminal Slope of a Semi-logarithmic Plasma Concentration-time Curve (t½λz) for Part A - Amorphous and Crystalline Suspension
Description: To assess Rate and extent of absorption of AZD5718 by assessment of the half-life associated with terminal slope of a semi-logarithmic plasma concentration-time curve (t½λz) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 11.90 (5.063) [1.00 to 5.98] | 13.14 (4.684) [1.00 to 2.98] | 13.30 (4.357) [0.50 to 3.03] | 14.62 (5.361) [0.52 to 1.00] | 11.62 (2.198) [0.98 to 2.00] | 10.41 (1.851) [1.00 to 2.00] | 19.97 (6.763) [1.00 to 4.00] | 14.18 (2.653) [1.00 to 5.98]

11. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Half-life Associated With Terminal Slope of a Semi-logarithmic Plasma Concentration-time Curve (t½λz) for Part B - Amorphous Suspension
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of the half-life associated with terminal slope of a semi-logarithmic plasma concentration-time curve (t½λz) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours
  Day 1 -From sampling time to 24 hrs; not true t½λz | 7.450 (0.8084) | 5.489 (1.168) | 5.920 (0.5085) | 6.799 (2.036)
  Day 10 | 11.65 (0.7718) | 11.29 (1.432) | 9.156 (1.014) | 10.23 (3.144)

12. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC (CL/F) for Part A - Amorphous and Crystalline Suspension
Description: To assess rate and extent of absorption of AZD5718 by assessment of the apparent total body clearance after extravascular administration estimated as dose divided by AUC (CL/F) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters/Hours
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters/Hours | 157.3 (60.18) [1.00 to 5.98] | 155.5 (22.31) [1.00 to 2.98] | 168.1 (74.10) [0.50 to 3.03] | 80.84 (18.41) [0.52 to 1.00] | 76.30 (29.08) [0.98 to 2.00] | 78.88 (31.04) [1.00 to 2.00] | 324.5 (77.99) [1.00 to 4.00] | 714.6 (292.2) [1.00 to 5.98]

13. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC (CL/F) for Part B - Amorphous Suspension
Description: To assess rate and extent of absorption of AZD5718 by assessment of the Rate and extent of absorption of AZD5718 by assessment of CL/F estimated as dose divided by AUC (for Day 1 only) and dose divided by AUCτ on Day 10 following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B)
Time Frame: Day 1 and Day 10 of Part B
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/Hour
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter/Hour
  Day 1 | 126.6 (31.39) | 112.2 (45.10) | 77.96 (24.80) | 85.85 (36.98)
  Day 10 | 99.85 (26.40) | 85.06 (35.38) | 65.65 (20.14) | 63.07 (28.39)

14. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) for Part A - Amorphous and Crystalline Suspension
Description: To assess rate and extent of absorption of AZD5718 by assessment of the apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: At post-dose (Days 1 to 3); 0.5, 1, 2, 3, 4, 6, 8, 24, 36 and 48 hours post-dose and folow up (Day 4 - 72 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liters | 2608 (447.6) [1.00 to 5.98] | 2940 (1063) [1.00 to 2.98] | 3490 (2433) [0.50 to 3.03] | 1770 (992.9) [0.52 to 1.00] | 1264 (446.6) [0.98 to 2.00] | 1189 (538.9) [1.00 to 2.00] | 8801 (2072) [1.00 to 4.00] | 14630 (5751) [1.00 to 5.98]

15. Secondary Outcome: To Evaluate the Relative Bioavailability Between the Amorphous and Crystalline Form of AZD5718 (Part A) by Assessment of AUC for Part A - Amorphous and Crystalline Suspension
Description: To assess the relative bioavailability by AUC between the cohort receiving the crystalline suspension and the corresponding data from the cohort receiving the same dose of the amorphous suspension (Part A only). Crystalline suspension was compared to the reference amorphous suspension.
  Note: Geometric mean ratios for crystalline/amorphous suspensions were calculated
Time Frame: At post-dose (Days 1 to 3); 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, and 48 hours post-dose and folow up (Day 4 - 72 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: h*nmol/L
Groups:
- 100 mg - AZD5718: Participants received single dose of oral suspension of AZD5718 100 mg in amorphous/crystalline state
- 300 mg - AZD5718: Participants received single dose of oral suspension of AZD5718 300 mg in amorphous/crystalline state
Arm/Group | 100 mg - AZD5718 | 300 mg - AZD5718
Number analyzed (Participants) | 6 | 6
h*nmol/L | 49.1 (2433) [34.0 to 70.7] | 11.9 (992.9) [8.38 to 16.9]

16. Secondary Outcome: To Evaluate the Relative Bioavailability Between the Amorphous and Crystalline Form of AZD5718 (Part A) by Assessment of Cmax for Part A - Amorphous and Crystalline Suspension
Description: To assess the relative bioavailability by Cmax between the cohort receiving the crystalline suspension and the corresponding data from the cohort receiving the same dose of the amorphous suspension (Part A only). Crystalline suspension was compared to the reference amorphous suspension.
  Note: Geometric mean ratios for crystalline/amorphous suspensions were calculated
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Groups:
- 100 mg AZD5718: Participants received single dose of oral suspension of AZD5718 100 mg in amorphous/crystalline state
Arm/Group | 100 mg AZD5718 | 300 mg - AZD5718
Number analyzed (Participants) | 6 | 6
nmol/L | 32.1 (2433) [20.8 to 49.4] | 3.40 (992.9) [2.35 to 4.92]

17. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Accumulation Ratio for AUC(0-τ) (RAC AUC(0-τ)) for Part B - Amorphous Suspension
Description: To assess rate and extent of absorption of AZD5718 by assessment of the Rate and extent of absorption of AZD5718 by assessment of accumulation ratio for AUC(0-τ) (RAC AUC(0-τ)) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B) Accumulation ratio calculated as AUC0-τ Day 10/AUC0-τ Day 1 (first dose) for Part B under fasted condition and presented values for Day 10
Time Frame: Day 1 and Day 9 (Part B only)
Population: as for outcome 2
Measure: Mean (Full Range); unit: Ratio
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio | 1.368 [1.13 to 1.57] | 1.387 [1.02 to 1.56] | 1.253 [0.848 to 1.48] | 1.444 [1.19 to 1.92]

18. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Accumulation Ratio for Cmax (RAC Cmax) for Part B (Amorphous Suspension) Under Fasted Condition
Description: To assess the rate and extent of absorption of AZD5718 by evaluation of accumulation ratio for Cmax (RAC Cmax) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B). Accumulation ratio calculated as Cmax Day 10/Cmax Day 1 (first dose) for Part B under fasted condition.
Time Frame: Day 1 and Day 9 (Part B only)
Population: as for outcome 2
Measure: Mean (Full Range); unit: Ratio, no units
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio, no units | 1.368 [1.13 to 1.57] | 1.387 [1.02 to 1.56] | 1.253 [0.848 to 1.48] | 1.444 [1.19 to 1.92]

19. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Temporal Change Parameter in Systemic Exposure (TCP) for Part B (Amorphous Suspension) Under Fasted Condition
Description: To assess rate and extent of absorption of AZD5718 by assessment of the temporal change parameter in systemic exposure (TCP) following a single AZD5718 dose on Day 1 and multiple daily dosing on Days 9 or 10 under fasted conditions (Part B).
  TCP calculated as AUCτDay10/AUCDay 1 and presented values for Day 10
Time Frame: At Day 10 (Part B only)
Population: as for outcome 2
Measure: Mean (Full Range); unit: Ratio, no units
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio, no units | 1.280 [1.08 to 1.45] | 1.349 [1.01 to 1.50] | 1.211 [0.822 to 1.44] | 1.385 [1.12 to 1.88]

20. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Effect of Food Following Administration of 180 mg AZD5718 With Food (Part B Day 9) and Fasted (Part B Day 10)
Description: The effect of food was evaluated by the assessment of the PK parameter (Cmax) following multiple daily doses of 180 mg AZD5718 under fasted condition (Part B Day 10) and immediately following a high-fat breakfast (Part B Day 9)
Time Frame: At Day 9 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- 180mg-Part B (Amorphous Suspension) -Fed State (Day 9): Participants received multiple doses of oral suspension of AZD5718 60 mg in amorphous state in 6 cohorts under fed condition
- 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10): Participants received multiple doses of oral suspension of AZD5718 180 mg in amorphous state in 6 cohorts under fed condition
Arm/Group | 180mg-Part B (Amorphous Suspension) -Fed State (Day 9) | 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10)
Number analyzed (Participants) | 6 | 6
nmol/L | 349.8 (34.99) | 1243 (55.23)
Statistical Analysis 1: Comparison: 180mg-Part B (Amorphous Suspension) -Fed State (Day 9) vs 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10); Cmax; Test type: Superiority or Other; Ratio = 28.13, 90% CI 2-sided [20.98 to 37.73]

21. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Effect of Food Following Administration of 180 mg AZD5718 With Food (Part B Day 9) and Fasted (Part B Day 10)
Description: The effect of food was evaluated by the assessment of the PK parameter (AUC(0-t) following multiple daily doses of 180 mg AZD5718 under fasted condition (Part B Day 10) and immediately following a high-fat breakfast (Part B Day 9)
Time Frame: At Day 9 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | 180mg-Part B (Amorphous Suspension) -Fed State (Day 9) | 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10)
Number analyzed (Participants) | 6 | 6
h*nmol/L | 3312 (33.26) | 5128 (46.90)
Statistical Analysis 1: Comparison: 180mg-Part B (Amorphous Suspension) -Fed State (Day 9) vs 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10); AUC(0-τ); Test type: Superiority or Other; Ratio = 64.58, 90% CI 2-sided [54.34 to 76.74]

22. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of the Effect of Food Following Administration of 180 mg AZD5718 With Food (Part B Day 9) and Fasted (Part B Day 10)
Description: The effect of food was evaluated by the assessment of the PK parameter(tmax) following multiple daily doses of 180 mg AZD5718 under fasted condition (Part B Day 10) and immediately following a high-fat breakfast (Part B Day 9)
Time Frame: At Day 9 and Day 10 (Part B only)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 180mg-Part B (Amorphous Suspension) -Fed State (Day 9) | 180mg -Part B (Amorphous Suspension) -Fasted State (Day 10)
Number analyzed (Participants) | 6 | 6
Hours | 3.51 [2.00 to 6.02] | 1.00 [0.98 to 1.02]

23. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Cumulative Amount of Analyte Excreted at the Last Sampling Interval (CumAe0-24) Following a Single Administration of AZD5718 Amorphous and Crystalline Suspension (Part A)
Description: To assess urine PK parameter (CumAe0-24) after a single administration of AZD5718 Amorphous suspension in Part A
Time Frame: Part A pre-dose and pooled intervals up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol | 206.9 (125.0) | 439.8 (85.95) | 1030 (449.7) | 5960 (2027) | 13610 (3850) | 23600 (8577) | 292.4 (80.50) | 425.9 (190.2)

24. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Percentage of Dose Excreted Unchanged Into the Urine From 0 to 24 Hours (Cumfe0-24) Following a Single Administration of AZD5718 Amorphous and Crystalline Suspension (Part A)
Description: To assess urine PK parameter (Cumfe0-24) estimated by dividing Ae(0-last) by dose after a single administration of AZD5718 Amorphous suspension in Part A
Time Frame: Part A pre-dose and pooled intervals up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Dose Excreted
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of Dose Excreted | 0.3695 (0.2232) | 0.3927 (0.07675) | 0.4598 (0.2008) | 0.8870 (0.3017) | 1.013 (0.2865) | 0.8781 (0.3191) | 0.1306 (0.03594) | 0.06339 (0.02831)

25. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Renal Clearance (CLR) Following a Single Administration of AZD5718 Amorphous and Crystalline Suspension (Part A)
Description: To assess the urine PK parameter (CLR) after a single administration of AZD5718 Amorphous suspension in Part A
Time Frame: Part A pre-dose and pooled intervals up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liter/hour | 0.7241 (0.2640) | 0.6221 (0.09344) | 0.6782 (1.599) | 0.6860 (0.1634) | 0.7093 (0.1118) | 0.6206 (0.07438) | 0.4502 (0.1043) | 0.4312 (0.07115)

26. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Cumulative Amount of Analyte Excreted From 0 to 24 Hours (CumAe0-24) Following a Multiple Daily Doses Administration of AZD5718 Amorphous Suspension (Part B Day 9)
Description: To assess the urine PK parameter (CumAe0-24) after a single administration of AZD5718 Amorphous suspension in Part B Day 9
Time Frame: Part B only, Day 9 at pooled 3 hour intervals until 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
nmol | 953.0 (253.2) | 2219 (612.0) | 13720 (612.0) | 18920 (6717)

27. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Percentage of Dose Excreted Unchanged Into the Urine From 0 to 24 Hours (Cumfe0-24) Following a Multiple Daily Doses Administration of AZD5718 Amorphous Suspension (Part B Day 9)
Description: To assess urine PK parameter (Cumfe0-24) estimated by dividing Ae(0-last) by dose after a single administration of AZD5718 Amorphous suspension in Part B Day 9
Time Frame: Part B only, Day 9 at pooled 3 hour intervals until 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Dose Excreted
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Dose Excreted | 0.7092 (0.1884) | 0.5504 (0.1518) | 1.702 (0.2911) | 1.408 (0.4999)

28. Secondary Outcome: Rate and Extent of Absorption of AZD5718 by Assessment of Renal Clearance (CLR) Following a Multiple Daily Doses Administration of AZD5718 Amorphous Suspension (Part B Day 9)
Description: To assess the urine PK parameter (CLR) after a single administration of AZD5718 Amorphous suspension in Part B Day 9
Time Frame: Part B only, Day 9 at pooled 3 hour intervals until 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter/hour | 0.6490 (0.1029) | 0.7172 (0.07593) | 0.9831 (0.04645) | 0.7368 (0.1654)

29. Secondary Outcome: Pharmacodynamic Analysis by ex Vivo Stimulation of Leukotriene B4 (LTB4) Production Using Calcium Ionophore for Part A -Amorphous and Crystalline Suspension
Description: To assess the change from baseline in the ex vivo stimulated LTB4 production using calcium ionophore in venous blood samples following a single administration of AZD5718 Amorphous and Crystalline suspension (Part A only)
Time Frame: Admission to 0.5, 1, 2, 3, 4, 6, 8, 24, 36 and 48 hours post-dose (Part A only)
Population: All subjects who received at least 1 dose of AZD5718 or placebo and who had at least 1 pre-dose and one post-dose measurement of stimulated LTB4 and who had no major protocol deviations thought to impact on the analysis of the PD data.
Measure: Median (Full Range); unit: Nanogram/liter (ng/L)
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | Placebo - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension) | Placebo - Part A (Crystalline Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 4
Nanogram/liter (ng/L)
  0.5 hours post-dose | 1.03 [0.689 to 1.18] | 0.877 [0.741 to 1.13] | 0.560 [0.200 to 0.813] | 0.000219 [0 to 0.00156] | 0.0000318 [0 to 0.000208] | 0 [0 to 0.0127] | 0.877 [0.496 to 2.60] | 0.781 [0.484 to 1.04] | 0.852 [0.532 to 1.23] | 0.934 [0.813 to 1.46]
  1.0 hours post-dose | 0.948 [0.787 to 1.19] | 0.553 [0.120 to 0.955] | 0.0213 [0.000343 to 0.332] | 0.0000451 [0 to 2.80] | 0 [0 to 0] | 0 [0 to 0] | 0.930 [0.414 to 2.52] | 0.497 [0.201 to 0.833] | 0.646 [0.363 to 1.02] | 0.833 [0.413 to 0.870]
  2.0 hours post-dose | 0.858 [0.150 to 1.20] | 0.124 [0.0144 to 0.543] | 0.000715 [0 to 0.0358] | 0 [0 to 0.000155] | 0 [0 to 0.000197] | 0 [0 to 0.0000955] | 0.943 [0.671 to 2.74] | 0.245 [0.0193 to 0.591] | 0.292 [0.0161 to 1.34] | 0.841 [0.372 to 1.34]
  3.0 hours post-dose | 0.672 [0.0415 to 1.34] | 0.0271 [0.00348 to 0.421] | 0.000165 [0 to 0.00218] | 0 [0 to 0.000217] | 0 [0 to 0] | 0 [0 to 0] | 0.965 [0.674 to 2.96] | 0.0449 [0.00161 to 0.134] | 0.0532 [0.000882 to 0.799] | 0.647 [0.449 to 1.36]
  4.0 hours post-dose | 0.616 [0.0234 to 0.925] | 0.0177 [0.00125 to 0.0904] | 0.000304 [0 to 0.00338] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0.952 [0.772 to 2.01] | 0.0187 [0.000422 to 0.0594] | 0.0329 [0 to 0.394] | 0.635 [0.0922 to 1.26]
  6.0 hours post-dose | 0.443 [0.0274 to 1.17] | 0.00669 [0.00296 to 0.0307] | 0.000249 [0 to 0.000884] | 0 [0 to 0.000607] | 0 [0 to 0.000330] | 0 [0 to 0.000267] | 1.20 [0.883 to 4.01] | 0.0267 [0.00503 to 0.0888] | 0.00819 [0.000518 to 0.147] | 0.842 [0.337 to 1.66]
  8.0 hours post-dose | 0.415 [0.0357 to 1.08] | 0.0234 [0.00890 to 0.104] | 0.000518 [0 to 0.0114] | 0 [0 to 0.000708] | 0 [0 to 0.000646] | 0 [0 to 0.000148] | 1.41 [1.00 to 3.63] | 0.0634 [0.00861 to 0.162] | 0.00880 [0.000418 to 0.212] | 1.39 [0.873 to 2.01]
  12.0 hours post-dose | 0.889 [0.0612 to 1.40] | 0.334 [0.0635 to 0.621] | 0.0515 [0.000546 to 0.210] | 0.00116 [0 to 0.00213] | 0.000106 [0 to 0.000469] | 0 [0 to 0.000149] | 1.36 [0.843 to 3.79] | 0.247 [0.0854 to 0.381] | 0.188 [0.00673 to 0.794] | 1.50 [0.226 to 2.45]
  24.0 hours post-dose | 0.874 [0.581 to 1.55] | 0.470 [0.394 to 0.716] | 0.435 [0.111 to 0.702] | 0.0698 [0.00817 to 0.197] | 0.00100 [0.000480 to 0.0135] | 0 [0 to 0.000308] | 1.04 [0.611 to 3.12] | 0.472 [0.249 to 0.747] | 0.369 [0.220 to 0.463] | 0.986 [0.910 to 2.00]
  36.0 hours post-dose | 1.91 [0.676 to 3.35] | 1.22 [0.620 to 2.15] | 0.813 [0.592 to 1.29] | 0.379 [0.205 to 1.23] | 0.0142 [0.00581 to 0.0405] | 0.00108 [0.000120 to 0.0643] | 1.70 [1.12 to 4.28] | 1.04 [0.831 to 1.47] | 1.04 [0.564 to 1.49] | 1.31 [1.08 to 2.40]
  48.0 hours post-dose | 1.48 [0.947 to 2.31] | 1.05 [0.808 to 1.74] | 0.739 [0.531 to 0.884] | 0.560 [0.411 to 1.40] | 0.290 [0.0790 to 0.484] | 0.0632 [0.000720 to 0.211] | 1.23 [0.689 to 5.46] | 0.638 [0.482 to 0.918] | 0.940 [0.512 to 1.29] | 0.893 [0.687 to 1.68]

30. Secondary Outcome: Pharmacodynamic Analysis by ex Vivo Stimulation of LTB4 Production Using Calcium Ionophore for Part B - Amorphous Suspension
Description: To assess the change from baseline in the ex vivo stimulated LTB4 production using calcium ionophore in venous blood samples following multiple administration of AZD5718 Amorphous suspension (Part B only)
Time Frame: Admission, predose and 0.5, 1, 2, 3, 4, 6, 8, 24, 36 and 48 hours post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: Nanogram/liter (ng/L)
Arm/Group | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension) | Placebo - Part B (Amorphous Suspension)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Nanogram/liter (ng/L)
  Day 1, 12 hours post-dose | 0.116 [0.00815 to 0.915] | 0.00171 [0.000244 to 0.0284] | 0.0000984 [0 to 0.000903] | 0 [0 to 0.000128] | 1.49 [1.11 to 2.55]
  Day 2, pre-dose | 0.654 [0.305 to 1.49] | 0.434 [0.121 to 0.816] | 0.00350 [0.00162 to 0.0440] | 0.000771 [0 to 0.00902] | 1.01 [0.510 to 1.80]
  Day 3, pre-dose | 0.557 [0.147 to 1.24] | 0.203 [0.0116 to 0.561] | 0.00609 [0.00131 to 0.0969] | 0.000893 [0 to 0.00343] | 1.10 [0.743 to 1.67]
  Day 4, pre-dose | 0.731 [0.230 to 1.54] | 0.294 [0.00887 to 1.61] | 0.00328 [0.000204 to 0.0229] | 0.000152 [0 to 0.00191] | 0.950 [0.787 to 2.05]
  Day 5, pre-dose | 0.421 [0.350 to 1.03] | 0.159 [0.000491 to 0.842] | 0.00467 [0.0000985 to 0.0498] | 0 [0 to 0.00110] | 0.893 [0.591 to 1.55]
  Day 6, pre-dose | 0.472 [0.148 to 1.29] | 0.227 [0.0148 to 2.18] | 0.00242 [0.000461 to 0.0226] | 0.000158 [0 to 0.00126] | 0.895 [0.488 to 1.35]
  Day 7, pre-dose | 0.511 [0.134 to 0.907] | 0.376 [0.00763 to 2.04] | 0.00210 [0.000188 to 0.0527] | 0.000195 [0 to 0.00420] | 1.05 [0.791 to 1.39]
  Day 8, pre-dose | 0.583 [0.170 to 0.962] | 0.134 [0.00223 to 0.782] | 0.00187 [0.000169 to 0.0255] | 0.000342 [0 to 0.00156] | 0.904 [0.625 to 1.44]
  Day 9, pre-dose | 0.288 [0.114 to 0.408] | 0.0360 [0.00731 to 0.274] | 0.00171 [0 to 0.00622] | 0.000130 [0 to 0.000597] | 0.661 [0.518 to 1.51]
  Day 10, pre-dose | 0.164 [0.0557 to 0.432] | 0.0266 [0.00483 to 0.153] | 0.000908 [0 to 0.00357] | 0 [0 to 0.000368] | 0.982 [0.292 to 1.37]
  Day 10, 2 hours post-dose | 0 [0 to 0.00153] | 0.000198 [0 to 0.00109] | 0 [0 to 0.000371] | 0 [0 to 0.000123] | 0.812 [0.270 to 1.36]
  Day 10, 6 hours post-dose | 0.000109 [0 to 0.000387] | 0.0000944 [0 to 0.000606] | 0 [0 to 0.000359] | 0 [0 to 0] | 0.921 [0.407 to 1.43]
  Day 10, 12 hours post-dose | 0.0143 [0.00140 to 0.0357] | 0.00247 [0 to 0.00772] | 0 [0 to 0.000390] | 0 [0 to 0.00109] | 1.20 [0.289 to 2.23]
  Day 11, 24 hours post-dose | 0.194 [0.105 to 0.355] | 0.0901 [0.00314 to 0.321] | 0.000426 [0 to 0.00130] | 0 [0 to 0.000279] | 1.20 [0.665 to 1.46]
  Day 12, 48 hours post-dose | 0.550 [0.193 to 1.10] | 0.906 [0.320 to 1.84] | 0.304 [0.0743 to 0.856] | 0.0583 [0.00295 to 0.813] | 1.05 [0.433 to 1.47]

ADVERSE EVENTS:
Time Frame: From screening to last follow-up visit (7-10 days after last dose), up to 6 weeks (Part A) and up to 8 weeks (Part B)
Description: All randomized subjects who received at least 1 dose of IMP and for whom any safety post dose-data were available were included in the safety analysis for the study. A treatment-emergent adverse event (TEAE) was defined as an AE with onset (start date/time) after the first dose of IMP.
Arm/Group | 25 mg - Part A (Amorphous Suspension) | 50 mg - Part A (Amorphous Suspension) | 100 mg - Part A (Amorphous Suspension) | 300 mg - Part A (Amorphous Suspension) | 600 mg - Part A (Amorphous Suspension) | 1200 mg - Part A (Amorphous Suspension) | Placebo - Part A (Amorphous Suspension) | 100 mg - Part A (Crystalline Suspension) | 300 mg - Part A (Crystalline Suspension) | Placebo - Part A (Crystalline Suspension) | 60 mg - Part B (Amorphous Suspension) | 180 mg - Part B (Amorphous Suspension) | 360 mg - Part B (Amorphous Suspension) | 600 mg - Part B (Amorphous Suspension) | Placebo - Part B (Amorphous Suspension)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 1/6 | 3/6 | 1/6 | 4/6 | 1/12 | 0/6 | 2/6 | 1/4 | 2/6 | 3/6 | 2/6 | 3/6 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg - Part A (Amorphous Suspension) (N=6) | 50 mg - Part A (Amorphous Suspension) (N=6) | 100 mg - Part A (Amorphous Suspension) (N=6) | 300 mg - Part A (Amorphous Suspension) (N=6) | 600 mg - Part A (Amorphous Suspension) (N=6) | 1200 mg - Part A (Amorphous Suspension) (N=6) | Placebo - Part A (Amorphous Suspension) (N=12) | 100 mg - Part A (Crystalline Suspension) (N=6) | 300 mg - Part A (Crystalline Suspension) (N=6) | Placebo - Part A (Crystalline Suspension) (N=4) | 60 mg - Part B (Amorphous Suspension) (N=6) | 180 mg - Part B (Amorphous Suspension) (N=6) | 360 mg - Part B (Amorphous Suspension) (N=6) | 600 mg - Part B (Amorphous Suspension) (N=6) | Placebo - Part B (Amorphous Suspension) (N=8)
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site reaction (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.